CLINICAL TRIAL: NCT05507970
Title: A First-in-Human, Single-Centre, Single Ascending Dose, Multiple Dose and Pilot Food Effect Study to Assess the Safety, Tolerability and Pharmacokinetics of MMV367 in Healthy Participants
Brief Title: First-in-Human Study to Assess the Safety, Tolerability and Pharmacokinetics of MMV367
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Quotient Sciences (Industry); Swiss BioQuant (Industry); Banook Group (Industry); The Doctors Laboratory Ltd (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMV_MMV367_21_01; 2022-000918-33 (EudraCT Number); ISRCTN17423851 (Registry Identifier: ISRCTN); 1005344 (Other: IRAS)
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Malaria,Falciparum
Keywords: Malaria; Healthy Volunteers
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Part 1 Single Ascending Dose Cohort A (Experimental): 100 mg MMV367, oral solution, fasted,
  Interventions: Drug: MMV367
- Part 1 Single Ascending Dose Cohort B (Experimental): Single ascending dose to be determined after SAC (Safety Advisory Committee) review of previous cohort.
  Intervention: MMV367, oral solution, fasted
  Interventions: Drug: MMV367
- Part 1 Single Ascending Dose Cohort C (Experimental): Single ascending dose to be determined after SAC review of previous cohort.
  Intervention: MMV367, oral solution, fasted
  Interventions: Drug: MMV367
- Part 1 Single Ascending Dose Cohort D (Experimental): Single ascending dose to be determined after SAC review of previous cohort.
  Intervention: MMV367, oral solution, fasted
  Interventions: Drug: MMV367
- Part 1 Single Ascending Dose Cohort Placebo (Placebo Comparator): Single ascending dose to be determined after SAC review of previous cohort.
  Intervention: placebo, oral solution, fasted
  Interventions: Drug: Placebo
- Part 2 Food Effect Fed 440mg (Experimental): Open label, 2-period cross-over, randomized, food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV367 determined to be safe in Part 1.
  MMV367: Single dose dispersed in sterile water.
  Interventions: Drug: MMV367 (Fed 440mg)
- Part 3 Multiple Dose Cohort A (Experimental): Double-blinded, randomised, placebo-controlled, multiple-dose study.
  Intervention: MMV367 oral solution, fasted. Once daily for 3 days.
  Interventions: Drug: MMV367
- Part 3 Multiple Dose Cohort A Placebo (Placebo Comparator): Double-blinded, randomised, placebo-controlled, multiple-dose study.
  Intervention: placebo, oral solution, fasted. Once daily for 3 days
  Interventions: Drug: Placebo
- Part 2 Food Effect Fasted 440mg (Experimental): Open label, 2-period cross-over, randomized, food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV367 determined to be safe in Part 1.
  Interventions: Drug: MMV367 (Fasted 440mg)

INTERVENTIONS:
Drug: MMV367 — Single dose dispersed in sterile water, fasted.
  Arms: Part 1 Single Ascending Dose Cohort A; Part 1 Single Ascending Dose Cohort B; Part 1 Single Ascending Dose Cohort C; Part 1 Single Ascending Dose Cohort D
Drug: Placebo — Single Dose dispersed in sterile water, fasted.
  Arms: Part 1 Single Ascending Dose Cohort Placebo
Drug: MMV367 (Fed 440mg) — Single dose dispersed in sterile water with a high fat meal.
  Other Names: Food Effect
  Arms: Part 2 Food Effect Fed 440mg
Drug: MMV367 — Single dose dispersed in sterile water, fasted, administered for 3 consecutive days.
  Other Names: Multiple dose
  Arms: Part 3 Multiple Dose Cohort A
Drug: Placebo — Single dose dispersed in sterile water, fasted, administered for 3 consecutive days.
  Other Names: Multiple dose
  Arms: Part 3 Multiple Dose Cohort A Placebo
Drug: MMV367 (Fasted 440mg) — Single dose dispersed in sterile water fasted.
  Other Names: Fasted
  Arms: Part 2 Food Effect Fasted 440mg

SUMMARY:
This three-part, first-in-human, healthy volunteer study aims to assess the safety and tolerability of the test medicine as well as how it is taken up by the body when given as single and multiple doses. The effect of food on the test medicine will also be investigated.

In Part 1, up to 40 volunteers will be split into up to 5 groups and will receive single oral doses of the test medicine or dummy medicine (placebo), at different dose levels.

In Part 2, up to 8 volunteers will receive one oral dose of the test medicine in the fed state and one oral dose in the fasted state.

In Part 3, up to 24 volunteers will be split into up to 3 groups and will receive single oral daily doses of the test medicine or placebo for 3 consecutive days.

Volunteers' blood and urine will be taken throughout the study for analysis of the test medicine and for their safety. In Part 1 and Part 3, volunteers will be discharged from the clinical unit 4 days after the final dose of the test medicine and will return to the clinical unit on two occasions for safety assessments to be performed. In Part 2, volunteers will be discharged from the clinical unit 4 days after the final dose of the test medicine and will return to the clinical unit on a single occasion for safety assessments to be performed. Volunteers are expected to be involved in this study for approximately 6 weeks for all study parts, from screening to the final return visit.

DETAILED DESCRIPTION:
Part 1 will be a double-blinded, randomised, placebo-controlled, single ascending dose (SAD) study, which will comprise up to 5 fasted cohorts (Cohorts 1A to 1E; Cohort 1E will be optional), with 8 participants in each cohort. Participants will be randomly assigned to receive a single oral dose of either active IMP (investigational medicinal product) (6 participants) or placebo (2 participants) to assess its safety, tolerability and PK (pharmacokinetic) profile. Each participant will take part in one cohort. Cohort A dose is 100mg. Doses for cohorts B to E will be determined following a blinded interim review of the safety, tolerability and PK data after each cohort, prior to the dose decision for subsequent cohorts.

Part 2 will be an open-label, randomised, balanced two-period crossover, food effect evaluation. It is planned to enrol 8 participants. In Period 1, participants will be randomised to 1 of 2 treatment sequences. If a participant is randomised to receive MMV367 in the fasted state in Period 1, they will receive MMV367 in the fed state in Period 2 and vice versa. The dose administered in Part 2 will be determined once predicted human therapeutic concentrations of MMV367 and a safe exposure window has been established in Part 1.

Part 3 will be a double-blinded, randomised, placebo-controlled, multiple-dose study. A total of 8 participants per cohort (A-C) will receive once-daily doses of MMV367 (6 participants) or placebo (2 participants) for 3 days, in the fasted state, to assess safety, tolerability and PK profile of multiple dosing. Cohorts 3B and 3C are optional and may proceed after a review of the safety and PK data. The dose(s) administered in Part 3 will be determined after review of the data from Part 1.

Parts 1 and 3 will follow a sentinel dosing design. For each of the three parts, participants will be screened within 28 days prior to first admission to the clinical unit on the morning of Day -1.

Part 1: In each cohort, participants will be dosed on Day 1 and will remain resident in the clinical unit until discharge on Day 5. They will attend the clinical unit for a return visit on Day 7 and again on Day 15 for end of study assessments.

Part 2: Participants will be dosed on Day 1 (Period 1 dose) and on Day 8 (Period 2 dose) and will remain resident in the clinical unit until discharge on Day 12. They will attend the clinical unit on Day 14 for end of study assessments. Based on emerging PK data from Part 1, the washout period between the Period 1 and Period 2 doses may be extended.

Part 3: Participants will receive a single dose on Days 1, 2 and 3 and will remain resident in the clinical unit until discharge on Day 7. They will attend the clinical unit for a return visit on Day 9 and again on Day 17 for end of study assessments.

For all parts, blood samples will be collected at regular intervals for PK analysis and safety from Day 1 to discharge from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent
2. Must be willing and able to communicate and participate in the whole study Demographics and Contraception
3. Aged 18 to 55 years inclusive at the time of signing informed consent
4. Must agree to adhere to the contraception requirements defined in Section 9.4 Baseline characteristics
5. Healthy males or non-pregnant, non-lactating healthy females.
6. Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening
7. Weight ≥50 kg at screening

Exclusion Criteria:

* Medical/Surgical History and Mental Health

  1. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
  2. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
  3. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
  4. Blood pressure (supine) at screening or admission outside the range of 90 to 140 mmHg systolic or 50 to 90 mmHg diastolic; and pulse rate outside the range of 45 to 100 bpm, unless deemed not clinically significant by the investigator
  5. A decrease of SBP (systolic blood Pressure) ≥20 mmHg after 3 min standing and/or a decrease of DBP (diastolic blood Pressure)

     ≥10 mmHg after 3 min standing, at screening
  6. History or presence of known structural cardiac abnormalities, family history of long QT (measured from the beginning of the QRS complex to the end of the T-wave) syndrome, cardiac syncope or recurrent, idiopathic syncope, exercise related clinically significant cardiac events. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QT interval changes
  7. Presence of sinus node dysfunction, clinically significant PR interval prolongation (>210 msec), intermittent second- or third-degree atrioventricular block, complete bundle branch block, sustained cardiac arrhythmias including (but not limited to) atrial fibrillation or supraventricular tachycardia; any symptomatic arrhythmia with the exception of isolated extra systoles, abnormal T wave morphology which may impact on the QT/QTc assessment, or QTcF >450 msec. Participants with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the sponsor's medical monitor and the investigator
  8. Participants with a history of cholecystectomy or gall stones
  9. Participants with conditions that affect their ability to smell or taste (Part 1 only) including, but not limited to mouth ulcers, gum disease, nasal surgery and smell and/or taste disorders (e.g. dysosmia, dysgeusia, respiratory and/or sinus infection or cold) Physical Examination
  10. Participants who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening Diagnostic assessments
  11. Evidence of current SARS-CoV-2 infection (severe acute respiratory syndrome)
  12. Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1 of protocol). Participants with Gilbert's Syndrome are not allowed.
  13. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) 1 and 2 antibody results
  14. Females who are pregnant or lactating (all female participants must have a negative highly sensitive serum pregnancy test at screening and a negative urine pregnancy test at admission) Prior Study Participation
  15. Participants who have received any IMP in a clinical research study within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer
  16. Participants who have previously been administered IMP in this study. Participants who have taken part in Part 1 are not permitted to take part in Parts 2 and 3 and participants who have taken part in Part 2 are not permitted to take part in Part 3
  17. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood Prior and Concomitant Medication
  18. Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day, hormonal contraception or HRT) in the 14 days before first IMP administration (see Section 11.4)
  19. Participants who have received a COVID-19 vaccine within 7 days before first IMP administration Lifestyle Characteristics
  20. History of any drug or alcohol abuse in the past 2 years
  21. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
  22. A confirmed positive alcohol breath test at screening or admission
  23. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
  24. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
  25. Confirmed positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1)
  26. Participant with a vegan or vegetarian diet (Part 2 only) Other
  27. Male participants with pregnant or lactating partners
  28. A score of 20 or more on the Beck Depression Inventory (BDI-II), and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) [7].

      Note, individuals with a BDI-II score of 17-19 may be enrolled, at the discretion of the investigator, if they do not have a medical history of psychiatric conditions and their mental state is not considered to pose additional risk to the health of the individual or to the execution of the trial and interpretation of the data
  29. Participants who are, or are immediate family members of, a study site or sponsor employee
  30. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Single Ascending Dose Cohort A 100mg; Part 1 Single Ascending Dose Cohort B 300mg; Part 1 Single Ascending Dose Cohort C 750mg; Part 1 Single Ascending Dose Cohort D 1500mg: MMV367: Single dose dispersed in sterile water.
- Part 1 Placebo: Received 100mg, 300mg, 750mg or 1500mg placebo oral solution.
  Placebo: Single dose dispersed in sterile water.
- Part 2 Food Effect Fed/Fasted 440mg; Part 2 Food Effect Fasted/Fed 440mg: Open label, 2-period cross-over, randomized, food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV367 determined to be safe in Part 1.
  MMV367: Single dose dispersed in sterile water.
- Part 3 Multiple Dose Cohort A 400mgx3: Double-blinded, randomised, placebo-controlled, multiple-dose study.
  Intervention: MMV367 or placebo, oral solution, fasted. Once daily for 3 days.
  MMV367: Single dose dispersed in sterile water.
- Part 3 Placebo: Received 400mg x3 placebo oral solution
  Placebo: 1 400mg dose per day for 3 days, dispersed in sterile water.
Period: Part 1: 100mg
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 6 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: 300mg
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: 750mg
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 0 | 0 | 6 | 0 | 1 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: 1500mg
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: 440mg First Intervention (1 Day)
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: 440mg Washout (7 Days)
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Second Intervention (1 Day)
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Multiple Dose Study
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed/Fasted 440mg | Part 2 Food Effect Fasted/Fed 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Single Ascending Dose Cohort A: 100mg MMV367 oral solution, fasted. Single dose dispersed in sterile water.
- Part 1 Single Ascending Dose Cohort B: Single ascending dose determined after SAC review of previous cohort.
  Intervention: 300mg MMV367 single dose dispersed in sterile water, fasted
- Part 1 Single Ascending Dose Cohort C: Single ascending dose determined after SAC review of previous cohort.
  Intervention: 750mg MMV367 single dose dispersed in sterile water, fasted
- Part 1 Single Ascending Dose Cohort D: Single ascending dose determined after SAC review of previous cohort.
  Intervention: 1500mg MMV367 single dose dispersed in sterile water, fasted
- Part 1 Single Ascending Dose Placebo: Single ascending dose determined after SAC review of previous cohort.
  Intervention: placebo, oral solution, fasted
- Part 2 Food Effect Fed/Fasted: Open label, 2-period cross-over, randomized, food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV367 determined to be safe in Part 1.
  MMV367: 440mg dispersed in sterile water in fed and fasted states.
- Part 2 Food Effect Fasted/Fed: Open label, 2-period cross-over, randomized, food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV367 determined to be safe in Part 1.
- Part 3 Multiple Dose 400mg: Double-blinded, randomised, placebo-controlled, multiple-dose study.
  Intervention: MMV367 400mg, oral solution, fasted. Once daily for 3 days.
  MMV367 400mg: Single dose dispersed in sterile water.
- Part 3 Multiple Dose Placebo: Double-blinded, randomised, placebo-controlled, multiple-dose study.
  Intervention: 400mg placebo, oral solution, fasted. Once daily for 3 days.
  MMV367: Single dose dispersed in sterile water.
  Placebo: Single dose dispersed in sterile water.
- Total: Total of all reporting groups
Arm/Group | Part 1 Single Ascending Dose Cohort A | Part 1 Single Ascending Dose Cohort B | Part 1 Single Ascending Dose Cohort C | Part 1 Single Ascending Dose Cohort D | Part 1 Single Ascending Dose Placebo | Part 2 Food Effect Fed/Fasted | Part 2 Food Effect Fasted/Fed | Part 3 Multiple Dose 400mg | Part 3 Multiple Dose Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 4 | 4 | 6 | 2 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (9.96) | 35.2 (6.59) | 41.3 (10.65) | 36.3 (6.44) | 40.1 (10.59) | 37.3 (8.88) | 29.3 (6.18) | 30.7 (11.36) | 39.5 (3.54) | 37.2 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 1 | 5 | 0 | 1 | 3 | 1 | 17
  Male | 3 | 5 | 4 | 5 | 2 | 4 | 3 | 3 | 1 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 6 | 6 | 7 | 4 | 4 | 6 | 2 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 5 | 5 | 5 | 5 | 6 | 4 | 4 | 5 | 2 | 41
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 6 | 7 | 4 | 4 | 6 | 2 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent AEs (TEAEs): AEs that commence during/after the first dose of IMP or commence before first dose of IMP (i.e., a pre-dose AE or existing medical condition) but worsen in intensity during exposure to IMP.
Time Frame: Screening/day-28 to EoS (End of Study) visit (Day 15 in Part 1, Day 14 in part 2 and Day 17 in part 3). Up to a maximum of 6.5 weeks in total.
Population: The data from the fed/fasted and fasted/fed arms are combined and are presented as fed and fasted. No calculations across/between arms were performed.
Measure: Number; unit: Number of events
Groups:
- Part 1 Placebo: Placebo: Single dose dispersed in sterile water.
- Part 2 Food Effect Fasted 440mg: Open label, 2-period cross-over, randomized, food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV367 determined to be safe in Part 1.
  MMV367: Single dose dispersed in sterile water.
- Part 3 Placebo: Placebo: 1 dose per day for 3 days, dispersed in sterile water.
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Number of events
  TEAEs | 1 | 4 | 5 | 1 | 5 | 2 | 1 | 12 | 12
  Severe TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  IMP-related TEAE | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to participant withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Clinically Significant Physical Examination Findings
Description: In the targeted (symptom driven) physical examination, a physician will assess the participant; if the participant reports feeling unwell or has ongoing AEs, then the physician will examine the appropriate body system(s) if required.
Time Frame: Screening/day-28 to EoS visit (Day 15 in Part 1, Day 14 in part 2 and Day 17 in part 3). Up to a maximum of 6.5 weeks in total
Population: as for outcome 1
Measure: Number; unit: Clinically significant abnormal finding
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Clinically significant abnormal finding | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Changes From Baseline for Electrocardiograms (ECGs): RR Interval (The R-R Interval is the Distance Between Two Consecutive R Waves.)
Description: Clinically important changes in mean values from baseline (individual: Day 1, Pre-dose; mean: Day 1, mean of 3 pre-dose measurements) to any post-dose time point
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: Number of clinically important changes
Groups:
- Part 1 Placebo: Received single placebo dose in sterile water.
- Part 3 Multiple Dose Cohort A 400mgx3: MMV367 once daily for 3 days in sterile water.
- Part 3 Placebo: Received placebo once daily for 3 days in sterile water.
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Number of clinically important changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Changes From Baseline for Laboratory Safety Tests (Haematology, Biochemistry)
Description: Shifts from within the reference range at baseline to outside the reference range after dosing with IMP.
Time Frame: Screening/day-28 to EoS visit (Day 15 in Part 1, Day 14 in part 2, and Day 17 in part 3). Up to a maximum of 6.5 weeks in total
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 Placebo: Received single dose placebo in sterile water.
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Participants
  Lymphocytes follow-up | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes Pre-dose D3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes 96 hr post last dose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT 24 hr: number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 0 | 0 | 0 | 0
  ALT 24 hr | 0 | 0 | 2 | 0 | 0 |  |  |  |
  ALT 96 hr post last dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0
  ALT 96 hr post last dose |  |  |  |  |  | 3 | 0 |  |
  ALT end of Study: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0
  ALT end of Study |  |  |  |  |  | 2 | 0 |  |
  Creatine kinase 144 hr post dose (144 hr post last dose Part 3): number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 0 | 0 | 6 | 2
  Creatine kinase 144 hr post dose (144 hr post last dose Part 3) | 0 | 2 | 0 | 3 | 0 |  |  | 0 | 1
  Protein follow-up: number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 0 | 0 | 6 | 2
  Protein follow-up | 0 | 2 | 0 | 0 | 0 |  |  | 0 | 0
  Calcium 24 hr post dose: number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 0 | 0 | 0 | 0
  Calcium 24 hr post dose | 0 | 0 | 0 | 0 | 2 |  |  |  |
  Calcium follow-up: number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 0 | 0 | 0 | 0
  Calcium follow-up | 2 | 0 | 0 | 0 | 0 |  |  |  |
  Calcium 48 hr post last dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Calcium 48 hr post last dose |  |  |  |  |  |  |  | 0 | 1
  Haematocrit 48 hr post last dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Haematocrit 48 hr post last dose |  |  |  |  |  |  |  | 2 | 0
  Neutrophils 48 hr post last dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Neutrophils 48 hr post last dose |  |  |  |  |  |  |  | 0 | 1
  Alkaline phosphatase pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Alkaline phosphatase pre-dose |  |  |  |  |  |  |  | 0 | 1
  Alkaline phosphatase 96 hr post last dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Alkaline phosphatase 96 hr post last dose |  |  |  |  |  |  |  | 0 | 1

5. Primary Outcome: Number of Clinically Important Changes From Baseline for Respiratory Rate
Description: Clinically important changes in mean values from baseline (Day 1, Pre-dose) to any post-dose time point for any dose level of MMV367 or placebo.
Time Frame: Screening/day-28 to EoS visit (Day 15 in Part 1, Day 14 in part 2,and Day 17 in part 3). Up to a maximum of 6.5 weeks in total
Population: as for outcome 1
Measure: Number; unit: Number of clinically important changes
Groups:
- Part 3 Placebo: Received placebo once daily in sterile water for 3 days.
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Number of clinically important changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Clinically Important Changes in Heart Rate, Supine
Description: as for outcome 5
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Number of clinically important changes
Groups:
- Part 3 Multiple Dose Cohort A 400mgx3: Received MMV367 once daily for 3 days in sterile water.
- Part 3 Placebo: Received placebo in sterile water once daily for 3 days.
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Number of clinically important changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Clinically Important Changes in Heart Rate, Orthostatic
Description: as for outcome 5
Time Frame: Screening/day-28 to Day 7 in Part 1, Day 15 in Part 2, and Day 9 in Part 3, up to a maximum of 6 weeks in total
Population: as for outcome 1
Measure: Number; unit: Number of clinically important changes
Groups:
- Part 2 Food Effect Fed 440mg: Open label, 2-period cross-over, randomized, food effect study to provide preliminary information on the effect of a high-fat meal on the pharmacokinetics of a single-dose oral administration of MMV367 determined to be safe in Part 1.
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Number of clinically important changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Clinically Important Changes From Baseline for Blood Bressure in mmHg: Orthostatic
Description: as for outcome 5
Time Frame: Screening/day-28 to Day 7 in Part 1, Day 15 in Part 2, and Day 9 in Part 3, up to a maximum of 6 weeks in total
Population: as for outcome 1
Measure: Number; unit: Number of clinically important changes
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Number of clinically important changes
  Systolic Orthostatic Change (mmHg) 6 hr | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Diastolic Orthostatic Change (mmHg) 6 hr | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Systolic Orthostatic Change (mmHg) 12 hr | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Orthostatic Change (mmHg) 12 hr | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  All other timepoints | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Changes From Baseline For Electrocardiograms (ECGs): QTcF (Corrected QT Interval Using the Fridericia Formula)
Description: Number of Participants with Out of Range QTcF Values
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Participants
  Between 450 to 480 msec | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Between 480 and 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prolongation between 30 to 60 msec | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Prolongation greater than 60 msec | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Changes From Baseline for Electrocardiograms (ECGs): QTcB (Corrected QT Interval Using the Bazett's Formula)
Description: Number of Participants with Out of Range QTcB Values
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Participants
  QTcB interval increase between 30 to 60 msec 1 hr | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec 3 hr | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  QTcB interval increase between 30 to 60 msec 5 hr | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec 6 hr | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec 8 hr | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec 12 hr | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  QTcB interval increase between 30 to 60 msec 24 hr | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec 72 hr | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec 96 hr | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec 144 hr | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec Follow-up | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  QTcB interval increase between 30 to 60 msec End of Study | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  QTcB interval increase between 30 to 60 msec D2 12 hr | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  QTcB interval increase between 30 to 60 msec D3 8 hr | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  QTcB interval increase between 30 to 60 msec D4 36 hr | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  All other timepoints | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Clinically Important Changes From Baseline for Blood Pressure in mmHg: Supine
Description: as for outcome 5
Time Frame: Screening/day -28 to EoS visit (Day 15 in Part 1, Day 14 in part 2, and Day 17 in Part 3). Up to a maximum of 6.5 weeks in total.
Population: as for outcome 1
Measure: Number; unit: Number of clinically important changes
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 8 | 8 | 6 | 2
Number of clinically important changes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs will be monitored from the time the participant signs the ICF (Informed Consent Form) until the end of study visit.
Groups:
- Part 1 Placebo: Received 100mg, 300mg, 750mg or 1500mg placebo in sterile water.
- Part 3 Multiple Dose Cohort A 400mgx3: MMV367 400mg once daily for 3 days in sterile water.
- Part 3 Placebo: Received 400mg x3 placebo in sterile water.
Arm/Group | Part 1 Single Ascending Dose Cohort A 100mg | Part 1 Single Ascending Dose Cohort B 300mg | Part 1 Single Ascending Dose Cohort C 750mg | Part 1 Single Ascending Dose Cohort D 1500mg | Part 1 Placebo | Part 2 Food Effect Fed 440mg | Part 2 Food Effect Fasted 440mg | Part 3 Multiple Dose Cohort A 400mgx3 | Part 3 Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/8 | 0/8 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/8 | 0/8 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 1/6 | 3/6 | 2/6 | 1/6 | 2/7 | 2/8 | 1/8 | 4/6 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Single Ascending Dose Cohort A 100mg (N=6) | Part 1 Single Ascending Dose Cohort B 300mg (N=6) | Part 1 Single Ascending Dose Cohort C 750mg (N=6) | Part 1 Single Ascending Dose Cohort D 1500mg (N=6) | Part 1 Placebo (N=7) | Part 2 Food Effect Fed 440mg (N=8) | Part 2 Food Effect Fasted 440mg (N=8) | Part 3 Multiple Dose Cohort A 400mgx3 (N=6) | Part 3 Placebo (N=2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulance (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dental parathesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and remove information and/or data that may impair the Sponsor's ability to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05507970/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT05507970/SAP_001.pdf